CLINICAL TRIAL: NCT05257187
Title: Shortening the Duration of Labor: Can We Remove Transcervical Foley Catheters Earlier
Brief Title: Foley Catheter Induction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants due to COVID pandemic
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Melissa Lozano, Assistant Professor - Obstetrics, Gynecology and Reproductive Science, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-21-00129
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Labor Induction

STUDY DESIGN:
Intervention Model Description: The study team will randomize patients to one of the following two groups: foley balloon removal after 6 hours or foley balloon removal after 12 hours. All patients will receive simultaneous pitocin and foley balloon. The remainder of the induction course (i.e. rupture of membranes, etc.) will be left to the discretion of the obstetric provider. The study is intention-to-treat meaning that if the foley balloon falls out earlier than the 6 hour or the 12 hour mark, the patient will still be included in the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 6 hour foley catheter retention (Active Comparator): Patients will have the foley catheter in place for up to 6 hours starting from insertion time to removal. If the catheter falls out earlier than the 6 hour mark, the patient will still be included for analysis.
  Interventions: Device: Transcervical foley catheter
- 12 hour foley balloon retention (Placebo Comparator): Patients will have the foley catheter in place for up to 12 hours starting from insertion time to removal. If the catheter falls out earlier than the 12 hour mark, the patient will still be included for analysis.
  Interventions: Device: Transcervical foley catheter

INTERVENTIONS:
Device: Transcervical foley catheter — The foley catheter is inserted manually by an obstetric provider through the cervix and inflated with 60cc of saline. Once in the correct position, the catheter is inflated, which puts pressure on the cervix, allowing it to release hormones that soften the cervix and help the cervix to open. The foley catheter can be left in place up to 12 hours but typically will fall out when the cervix is dilated to 3-4 centimeters.

SUMMARY:
The foley catheter (single lumen balloon) is one of the most cost effective, readily available methods for cervical ripening to begin an induction of labor. It is most commonly used in conjunction with oxytocin, a medication given to induce contractions. However, there is no clear timeline for when to remove the foley catheter or how long foley catheters can be safely kept in place.

The study team's goal is to conduct a randomized controlled trial (RCT) in nulliparous and multiparous patients to determine the optimal length of time to retain foley catheters (single balloon) for induction of labor to achieve vaginal delivery while shortening the overall length of labor. Based on our power analysis, the study team plans to enroll a total of 356 patients (218 nulliparous patients and 138 multiparous patients) over the course of 18 months.

Then the study team will randomize patients to one of the following two groups: foley catheter removal after 6 hours or foley catheter removal after 12 hours. All patients will receive simultaneous pitocin and a foley catheter, and the remainder of the induction course (i.e. rupture of membranes, etc.) will be left to the discretion of the obstetric provider. The primary outcome will be time of foley catheter insertion to delivery. Secondary outcomes will be rates of cesarean delivery and obstetric/neonatal outcomes.

DETAILED DESCRIPTION:
The study team's goal is to conduct a randomized controlled trial in nulliparous and multiparous patients to determine the optimal length of time to retain foley catheters (single balloon) for induction of labor to achieve vaginal delivery while shortening the overall length of labor. The primary hypothesis is that removal of the single balloon foley catheter at 6 hours after insertion compared to removal at 12 hours results in no difference in time to delivery and does not increase the cesarean delivery rate for nulliparous patient or for multiparous patients.

Background Nearly one quarter of all deliveries at term, in developed countries, involve an induction of labor. When labor induction begins, a baseline cervical exam is performed to determine a Bishop score and whether cervical ripening is indicated with medications (e.g misoprostol) or mechanical methods (foley catheter single catheter or cook catheter double balloon). The literature suggests that foley catheters can be removed without waiting for spontaneous expulsion with no difference in the length of labor, but there is no clear timeline for when to remove the foley catheter or how long foley catheters can be safely kept in place. One RCT found that the time from Cook catheter insertion to delivery is shorter by 5.8 hours for nulliparous patients and by 4.7 hours for multiparous patients without worsening maternal or neonatal outcomes

.

A recent publication found similar results applicable to single balloon foley catheters. In that study, patients randomized to foley balloon removal at 6 hours had a statistically significant shorter insertion-to-delivery time by 5 hours compared to the 12-hour removal group with no increase in the cesarean delivery rate. Although this study was the first randomized controlled trial to compare the use of foley catheters for labor induction for up to 6 hours retention vs. 12 hours retention, the study was underpowered for multiparous patients. The researchers are hoping to contribute the knowledge gap about the optimal time to retain foley catheters particularly in multiparous patients.

Longer labors have been associated with an increased risk of a prolonged second stage, maternal fever, shoulder dystocia, and admission to a level 2 or 3 nursery. In the advent of the ARRIVE Trial, more patients are now undergoing induction of labor, so obstetric providers are incentivized to provide efficient and safe methods of labor induction that are effective at achieving vaginal delivery. The study team's goal is to conduct a randomized controlled trial in nulliparous and multiparous women to determine the optimal length of time to retain foley catheters (single balloon) for induction of labor to achieve vaginal delivery while shortening the overall length of labor.

At the institution (Mount Sinai West), the study team will use foley catheters instead of cook catheters and there is a trend towards waiting for spontaneous expulsion. The study team will collect demographic and pregnancy data about patients and determine if they meet inclusion criteria. Then the study team will randomize patients to one of the following two groups: foley catheter removal after 6 hours or foley catheter removal after 12 hours. All patients will receive simultaneous pitocin and foley catheter. The remainder of the induction course (i.e. rupture of membranes, etc.) will be left to the discretion of the obstetric provider.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 50 years old
* Bishop score of 6 or less
* Singleton pregnancies at 37 weeks or more
* Absence of labor or rupture of membranes.

Exclusion Criteria:

* COVID positive patients
* Previous history of cesarean delivery
* Ruptured membranes (the institutional policy states women cannot have foley catheters placed if membranes are ruptured)
* Documented labor on admission (will include only patients being induced)
* Fetal distress on admission (e.g. indication for induction of labor being category 2 tracing as these patients may have increased risk of cesarean delivery)
* Certain fetal anomalies (e.g. brain anomalies, abdominal wall or neural tube defects, fetal cardiac arrhythmias)
* Contraindication to vaginal delivery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-07 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Length of Labor | Day 1, at time of infant delivery
  Length of time from foley catheter insertion to delivery time in minutes at the time of infant delivery

SECONDARY OUTCOMES:
Number of Cesarean delivery | Day 1, at time of infant delivery
  Number of delivery by Cesarean delivery
Number of Maternal Intrapartum Fever | Day 1, at time of infant delivery
  Number of participants with intrapartum fever
Number of Participants that require Intrapartum antibiotic administration | Day 1, at time of infant delivery
  Number of Participants that require Intrapartum antibiotic administration
Number of Participants with Postpartum Hemorrhage | 6 Days Postpartum
  Number of participants who had postpartum hemorrhage
Number of NICU admission | 6 Days Postpartum
  The number of babies delivered by patients enrolled in the study who ended up admitted to the Neonatal Intensive Care Unity (NICU) for any amount of time
Number of neonatal participants with APGAR score <7 | Day 1, 5 minutes of infant delivery
  Number of neonatal participants with 5 minute APGAR <7. APGAR score range is from 0-10, with the higher scores indicating better health outcome.
Number of neonatal participants with hospital stay greater than 6 days | 6 Days Postpartum
  Number of neonatal participants with hospital stay greater than 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Lois Brustman, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Bleicher I, Dikopoltsev E, Kadour-Ferro E, Sammour R, Gonen R, Sagi S, Eshel A, Nussam L, Vitner D. Double-Balloon Device for 6 Compared With 12 Hours for Cervical Ripening: A Randomized Controlled Trial. Obstet Gynecol. 2020 May;135(5):1153-1160. doi: 10.1097/AOG.0000000000003804. PMID 32282603
- [Background] Lassey SC, Haber HR, Kanbergs A, Robinson JN, Little SE. Six versus twelve hours of single-balloon catheter placement with oxytocin administration for labor induction: a randomized controlled trial. Am J Obstet Gynecol. 2021 Jun;224(6):611.e1-611.e8. doi: 10.1016/j.ajog.2021.03.021. Epub 2021 Mar 23. PMID 33771496